CLINICAL TRIAL: NCT04723563
Title: INHALEd Unfractionated HEParin for the Treatment of Hospitalized Patients With COVID-19 Pneumonia
Brief Title: Nebulized Heparin for the Treatment of COVID-19
Acronym: INHALE-HEP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Frederick Health (Other)
Responsible Party: Principal Investigator, Thomas Smoot, PharmD, Primary Investigator, Frederick Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FHHep2121
Record Dates: First submitted 2021-01-22; First posted 2021-01-25 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Covid19; Pneumonia, Viral
Keywords: heparin; COVID-19
MeSH Terms: conditions — COVID-19; Pneumonia, Viral | interventions — Heparin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Nebulized Heparin (Experimental): Heparin 5,000 units/mL Dose: 25,000 units Frequency: Four times per day Duration: until hospital discharge
  Interventions: Drug: Heparin
- Placebo (Placebo Comparator): 0.9% Sodium Chloride Dose: 5 mL Frequency: Four times per day Duration: until hospital discharge
  Interventions: Drug: 0.9%sodium chloride

INTERVENTIONS:
Drug: Heparin — 25,000 units of unfractionated heparin nebulized 4 times daily for the duration of hospitalization
  Arms: Nebulized Heparin
Drug: 0.9%sodium chloride — 5 mL of 0.9% sodium chloride nebulized 4 times daily for the duration of hospitalization
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Randomized, placebo controlled study to determine if nebulized heparin may reduce the need for mechanical ventilation in hospitalized patients with the novel coronavirus, also known as COVID-19. This will be a part of a larger meta-trial.

DETAILED DESCRIPTION:
COVID-19 is a novel coronavirus that can cause severe and potentially fatal respiratory infections. COVID-19 has many similarities to previously seen coronaviruses, such as those that caused the Middle Eastern Respiratory Syndrome (MERS) that emerged in 2011 and the Severe Acute Respiratory Syndrome (SARS) in 2002-2003. Based on early reports, many patients may present with mild to moderate respiratory symptoms, but approximately 20% developed severe symptoms. These severe cases developed a multitude of life threatening complications, like acute lung injury (ALI), acute respiratory distress syndrome (ARDS), and shock.

An early investigation into the patients with severe presentations, revealed high levels of inflammatory cytokines like interleukin 2 (IL-2), interleukin 6 (IL-6), tumor necrosis factor alpha (TNF-α), and monocyte chemoattractant protein 1 (MCP-1). This upregulation of inflammatory cytokines, also referred to as a cytokine storm, is similar to the innate immune response triggered by the previous coronaviruses.5,6 The increased production of these cytokines is the expected anti-viral response of the innate immune system, which is trigged by viral RNA replication. Viral replication triggers downstream inflammatory signaling cascades like NF-κB and IRF3 leading to increased neutrophil and monocyte-macrophages infiltrating the tissue. While effective against viral infection, this process is also believed to be responsible for the development of the significant respiratory complications associated with COVID-19.

ALI and ARDS are not unique to COVID-19 and develop with many viral respiratory infections. Several therapeutic strategies have been evaluated in ALI and ARDS and demonstrated benefit outside of the current pandemic. Heparin, a commonly used anticoagulant, has been shown to exhibit anti-inflammatory properties within the respiratory system. An in vitro study of heparin in a pulmonary cell model of ALI found that heparin significantly inhibited the NF-κB pathway. This inhibition led to a reduced levels of IL-6 and TNF-α in human alveolar macrophages exposed to an E. coli lipopolysaccharide to simulate inflammatory ALI. Additionally, heparin significantly reduced IL-6, TNF-α, and MCP-1 in human alveolar type II cell models. No increases in necrosis or apoptosis were observed.

In addition to these immunomodulation effects, heparin is primarily an anticoagulant and systemic administration carries a risk of bleeding. Due to this, several investigations were conducted in animal models and in humans to determine if administering the heparin via nebulization could take advantage of the immunomodulation, without increasing the risk of bleeding. Nebulized heparin was studied in a rat model of ARDS and was observed to attenuate ALI through reduction of pro-coagulant and pro-inflammatory pathways. Significant reductions in IL-6 and TNF-α were observed. Additionally, reductions in the expression of NF-κB were observed in the alveolar macrophages.

Several clinical investigations in humans with ARDS have also been completed. In a randomized, placebo controlled study of 60 patients with severe ARDS, patients were randomized to nebulized heparin, streptokinase and placebo. Patients in the heparin group received 10,000 units via nebulizer every 4 hours and had significant improvements in their ARDS by day 8. No effect on systemic coagulation markers like APTT and INR were observed. Additionally, no major bleeding events or blood transfusions were observed. A second, randomized placebo controlled trial of 50 patients requiring more than 48 hours of mechanical ventilation was conducted to determine the possible benefit of nebulized heparin. Patients with ALI that received nebulized heparin had a significant reduction in the time on the ventilator as compared to placebo. Patients that received heparin had higher APTT values than those that received placebo, but no significant bleeding events occurred. This study utilized a heparin dose of 25,000 units every 4 hours, which may explain the difference between the laboratory effects in the two human studies.

Heparin has demonstrated the ability to reduce the inflammatory cytokines believed to be responsible for the development of ALI and ARDS in COVID-19 and it may prove to be beneficial in this patient population. When administered via nebulization, no adverse effects were observed in the previously conducted studies and may provide a safe therapeutic option to improve the outcomes of patients with COVID-19 related ALI and ARDS.

This study will be a randomized, double-blind, placebo controlled trial to determine if nebulized heparin administered for the duration of hospitalization will reduce the need for mechanical ventilation and the overall length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the hospital
* There is a PCR positive sample for SARS-CoV-2 within the past 21 days. The sample can be a nasal orpharyngeal swab, sputum, tracheal aspirate, bronchoalveolar lavage, or another sample from the patient
* Modified Ordinal Clinical Scale for COVID-19 of 3-5

Exclusion Criteria:

* Intubated and on mechanical ventilation, or requiring immediate intubation as per the treating clinician's assessment
* Heparin allergy or heparin-induced thrombocytopaenia
* APTT > 120 seconds, not due to anticoagulant therapy and does not correct with administration of fresh frozen plasma
* Platelet count < 20 x 109 per L
* Pulmonary bleeding or uncontrolled bleeding
* Pregnant or might be pregnant
* Acute brain injury that may result in long-term disability
* Myopathy, spinal cord injury, or nerve injury or disease with a likely prolonged incapacity to breathe independently e.g. Guillain-Barre syndrome
* Treatment limitations in place, i.e. not for intubation, not for ICU admission
* Death is imminent or inevitable within 24 hours
* Clinician objection
* Refusal of participant (person responsible) consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2021-08-23 (Actual)

PRIMARY OUTCOMES:
Need for mechanical ventilation at day 28 | 28 days
  proportion of patients needed mechanical ventilation by day 28

SECONDARY OUTCOMES:
Hospital length of stay | 60 days
  Days of hospital admission
Average daily SaO2/FiO2 | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Frederick Health Hospital, Frederick, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Prompetchara E, Ketloy C, Palaga T. Immune responses in COVID-19 and potential vaccines: Lessons learned from SARS and MERS epidemic. Asian Pac J Allergy Immunol. 2020 Mar;38(1):1-9. doi: 10.12932/AP-200220-0772. PMID 32105090
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Liu B, Li M, Zhou Z, Guan X, Xiang Y. Can we use interleukin-6 (IL-6) blockade for coronavirus disease 2019 (COVID-19)-induced cytokine release syndrome (CRS)? J Autoimmun. 2020 Jul;111:102452. doi: 10.1016/j.jaut.2020.102452. Epub 2020 Apr 10. PMID 32291137
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Mahallawi WH, Khabour OF, Zhang Q, Makhdoum HM, Suliman BA. MERS-CoV infection in humans is associated with a pro-inflammatory Th1 and Th17 cytokine profile. Cytokine. 2018 Apr;104:8-13. doi: 10.1016/j.cyto.2018.01.025. Epub 2018 Feb 2. PMID 29414327
- [Background] Wong CK, Lam CW, Wu AK, Ip WK, Lee NL, Chan IH, Lit LC, Hui DS, Chan MH, Chung SS, Sung JJ. Plasma inflammatory cytokines and chemokines in severe acute respiratory syndrome. Clin Exp Immunol. 2004 Apr;136(1):95-103. doi: 10.1111/j.1365-2249.2004.02415.x. PMID 15030519
- [Background] Perlman S, Dandekar AA. Immunopathogenesis of coronavirus infections: implications for SARS. Nat Rev Immunol. 2005 Dec;5(12):917-27. doi: 10.1038/nri1732. PMID 16322745
- [Background] Darden DB, Hawkins RB, Larson SD, Iovine NM, Prough DS, Efron PA. The Clinical Presentation and Immunology of Viral Pneumonia and Implications for Management of Coronavirus Disease 2019. Crit Care Explor. 2020 Apr 29;2(4):e0109. doi: 10.1097/CCE.0000000000000109. eCollection 2020 Apr. PMID 32426751
- [Background] Camprubi-Rimblas M, Guillamat-Prats R, Lebouvier T, Bringue J, Chimenti L, Iglesias M, Obiols C, Tijero J, Blanch L, Artigas A. Role of heparin in pulmonary cell populations in an in-vitro model of acute lung injury. Respir Res. 2017 May 10;18(1):89. doi: 10.1186/s12931-017-0572-3. PMID 28486961
- [Background] Chimenti L, Camprubi-Rimblas M, Guillamat-Prats R, Gomez MN, Tijero J, Blanch L, Artigas A. Nebulized Heparin Attenuates Pulmonary Coagulopathy and Inflammation through Alveolar Macrophages in a Rat Model of Acute Lung Injury. Thromb Haemost. 2017 Nov;117(11):2125-2134. doi: 10.1160/TH17-05-0347. Epub 2017 Nov 30. PMID 29202212
- [Background] Abdelaal Ahmed Mahmoud A, Mahmoud HE, Mahran MA, Khaled M. Streptokinase Versus Unfractionated Heparin Nebulization in Patients With Severe Acute Respiratory Distress Syndrome (ARDS): A Randomized Controlled Trial With Observational Controls. J Cardiothorac Vasc Anesth. 2020 Feb;34(2):436-443. doi: 10.1053/j.jvca.2019.05.035. Epub 2019 May 27. PMID 31262641
- [Background] Dixon B, Schultz MJ, Smith R, Fink JB, Santamaria JD, Campbell DJ. Nebulized heparin is associated with fewer days of mechanical ventilation in critically ill patients: a randomized controlled trial. Crit Care. 2010;14(5):R180. doi: 10.1186/cc9286. Epub 2010 Oct 11. PMID 20937093
- [Background] van Haren FMP, Page C, Laffey JG, Artigas A, Camprubi-Rimblas M, Nunes Q, Smith R, Shute J, Carroll M, Tree J, Carroll M, Singh D, Wilkinson T, Dixon B. Nebulised heparin as a treatment for COVID-19: scientific rationale and a call for randomised evidence. Crit Care. 2020 Jul 22;24(1):454. doi: 10.1186/s13054-020-03148-2. PMID 32698853